CLINICAL TRIAL: NCT06363890
Title: Frequency and Etiology of Travelers' Diarrhea in Australian Adult Tourists Traveling to Southeast Asia
Brief Title: Etiology of Travelers' Diarrhea in Australian Tourists Traveling to Southeast Asia
Acronym: AusTD
Status: Recruiting | Type: Observational
Sponsor: Lumen Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TD02
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Travelers Diarrhea
Keywords: travelers diarrhea; australian; epidemiology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Australian travelers: 1200 Healthy Australian adult tourists traveling to Southeast Asia.
  Interventions: Diagnostic Test: TAQMan Array Card

INTERVENTIONS:
Diagnostic Test: TAQMan Array Card — Real time PCR test to detect diarrheal pathogens.

SUMMARY:
The study proposed here will determine the frequency and etiology of diarrhea in Australian adult tourists traveling to Southeast Asia, including Cambodia, Indonesia, Laos, Malaysia, Myanmar, the Philippines, Thailand, Timor-Leste, and Vietnam. The results from this study will inform the feasibility and design of subsequent clinical trials of travelers' diarrhea interventions in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged > 18 years residing in Australia.
* Planned travel for 14 to 28 days starting in the next 30 days to selected countries in Southeast Asia, including Cambodia, Indonesia, Laos, Malaysia, Myanmar, the Philippines, Thailand, Timor-Leste, and Vietnam.
* Willing to participate in the clinical study and available for all planned study activities through approximately 28 days post-travel.
* Access to a smartphone and mobile phone services while traveling (either by local SIM card, WiFi, or international roaming service on the individual's home-country mobile phone).

Exclusion Criteria:

* Unable or unwilling to provide adequate informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1200 Australian adult tourists traveling to Southeast Asia
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Characterize the frequency and etiology of travelers' diarrhea in this participant population of Australian adult tourists traveling to Southeast Asia. | 18 months
  Incidence of new episodes of self-reported diarrhea per 100 person-months of travel in enrolled participants.
  Among participants returning stool collection cards, compare the adjusted incidence of diarrhea attributed to specific etiologies.

CONTACTS AND LOCATIONS:
Locations (1):
- AK Clinical Research, Melbourne, Australia